CLINICAL TRIAL: NCT00842400
Title: A Phase I, Single-Center, Open-Label, Non-randomized, One-Sequence Crossover, Pharmacokinetic Interaction Study of the Combination Product VI-0521 (Phentermine Plus Topiramate) With Metformin, Sitagliptin or Probenecid in Healthy Subjects
Brief Title: A Drug Interaction Study of VI-0521 With Metformin, Sitagliptan and Probenecid in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wesley Day, VP Clinical, Vivus, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: OB-107
Record Dates: First submitted 2009-02-06; First posted 2009-02-12 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Metformin; Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Metformin, VI-0521, Sitagliptan, Probenecid — This trial is an open-label, non-randomized, one-sequence crossover study.
  * metformin 500 mg tablet twice daily on Days 1 to 5 and on Days 30 to 34
  * sitagliptan 100 mg tablet once daily on Days 6 to 10 and on Days 35 to 39
  * VI-0521 (phentermine/topiramate) capsule once daily each morning at 3.75/23 mg for 2 days (Days 11-12), 7.5/46 mg for 3 days (Days 13-15), 11.25/69 mg for 3 days (Days 16-18) and 15/92 mg for 21 days (Days 19-39)
  * 2 g (four 500 mg) probenecid tablets on Day 29.
  Other Names: VI-0521, Sitagliptan, Metformin, Probenecid

SUMMARY:
The purposes of this study are to:

* Find out how much of the study drugs are in the blood of healthy subjects after taking multiple doses of VI-0521, metformin and sitagliptan.
* Determine the effect of probenecid on the amount of VI-0521 in the blood of healthy subjects after taking multiple doses.
* Find out how much topiramate is in the semen of healthy male subjects after taking multiple doses.

DETAILED DESCRIPTION:
This trial is an open-label, non-randomized, one-sequence crossover study. All subjects will receive an oral dose of metformin 500 mg tablet twice daily on Days 1 to 5 and on Days 30 to 34; an oral dose of sitagliptin 100 mg tablet once daily on Days 6 to 10 and on Days 35 to 39 and a single oral dose of VI-0521 (phentermine/topiramate) capsule once daily each morning at 3.75/23 mg for 2 days (Days 11-12), 7.5/46 mg for 3 days (Days 13-15), 11.25/69 mg for 3 days (Days 16-18) and 15/92 mg for 21 days (Days 19-39) plus a single oral dose of 2 g (four 500 mg) probenecid tablets on Day 29.

Subjects will remain at the site for the duration of the study (from Day -1 to Day 40). Blood samples for the determination of metformin concentrations in plasma will be collected at 0 (pre-dose), 1, 2, 3, 4, 6, 8 and 12 hours after the morning administration of metformin or metformin plus VI-0521 on Days 5 and 34. Blood samples for the determination of sitagliptin concentrations in plasma will be collected at 0 (pre-dose), 1, 2, 3, 4, 5, 7, 10, 16 and 24 hours after the administration of sitagliptin or sitagliptin plus VI-0521 on Days 10 and 39. Blood samples for the determination of phentermine and topiramate concentrations in plasma will be collected at 0 (pre-dose), 1, 2, 3, 4, 5, 7, 10, 16 and 24 hours after the administration of the investigational product(s) on Days 28, 29, 34 and 39. Pre-dose blood samples for determination of the investigational drug concentrations in plasma will be taken in the morning on Days 4 and 33 for metformin; Days 9 and 38 for sitagliptin and Days 27, 33 and 38 for phentermine and topiramate. Semen samples for determination of topiramate concentrations will be collected on Day 28 between five and seven hours after VI-0521 administration in 8 male non-vasectomized subjects to obtain at least 6 evaluable subjects.

The primary endpoints of this study will be the PK parameters AUC0-τ and Cmax of phentermine, topiramate, sitagliptin and metformin.The secondary endpoint is the topiramate concentration in semen.

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of adult healthy males or females, 19-45 years of age; inclusive who are medically healthy with no clinically significant screening results.

Exclusion Criteria:

* Main exclusion criteria include a history or presence of significant cardiovascular, neurological, hematological, psychiatric, hepatic, gastrointestinal, pulmonary, endocrine, immunologic or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs or place the subjects at increased risk as determined by the Investigator; any clinically significant laboratory abnormalities as judged by the Investigator; any history of glaucoma, increased intraocular pressure, or medications to treat increased intraocular pressure; presence of cholelithiasis or cholecystitis within the last 6 months that has not been surgically treated with cholecystectomy; any history of a cardiovascular or cerebrovascular event; any active malignancy except basal cell carcinoma; systolic blood pressure > 150 mm Hg or diastolic blood pressure > 95 mm Hg at screening or at check-in (Two rechecks are allowed); positive drug/alcohol test at screening or check in; blood donation or significant blood loss within 56 days of dosing; plasma donation within 7 days of dosing. In female subjects, a positive pregnancy test at screening or check-in is exclusionary.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoints of this study will be the PK parameters AUC0-τ and Cmax of phentermine, topiramate, sitagliptin and metformin. | 40 days

SECONDARY OUTCOMES:
The secondary endpoint is the topiramate concentration in semen. | 40 days

CONTACTS AND LOCATIONS:
Overall Officials: Shiyin Yee, Study Director — VIVUS LLC
Locations (1):
- MDS Pharma Services, Phoenix, Arizona, United States